CLINICAL TRIAL: NCT00693836
Title: Resource for the Study of Lung Cancer Epidemiology in North Trent
Brief Title: Studying Patterns, Causes, and Control of Disease in Patients With Lung Cancer in the North Trent (England) Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research Centre at Weston Park Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRC-WPH-USMS-ReSoLuCENT; CDR0000589308 (Registry Identifier: PDQ (Physician Data Query)); EU-20826
Record Dates: First submitted 2008-06-06; First posted 2008-06-09 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-12

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Genetic Linkage; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: genetic linkage analysis
Genetic: loss of heterozygosity analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: biologic sample preservation procedure
Other: medical chart review
Other: questionnaire administration
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Gathering information about genetic and environmental factors from patients with lung cancer and their partners and first-degree relatives may help doctors learn more about the disease.

PURPOSE: This clinical trial is looking at the patterns, causes, and control of disease in patients with lung cancer in the North Trent (England) region.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish a resource bank of high quality genomic and plasma DNA and tumor and serum samples linked to clinical data obtained from detailed family history and lifestyle questionnaires from patients with lung cancer and from their partners and first-degree relatives for genetic epidemiology studies of lung cancer.

Secondary

* To study single nucleotide polymorphisms for candidate lung cancer susceptibility genes in genomic DNA samples from patients with lung cancer and from their partners and first-degree relatives.
* To study genetic changes of lung cancer in plasma DNA samples from patients with lung cancer and from their partners and first-degree relatives.

OUTLINE: This is a multicenter study.

Patients and their partners complete a detailed, interview-based questionnaire to assess their environmental risk factors for cancer. Information on past medical, social, occupational, and smoking history as well as family history, including any malignancies diagnosed and subsequent causes of death, is collected. First-degree relatives of patients complete an interview-based questionnaire about smoking, occupational, and cancer history. Relatives of patients' partners complete a telephone-administered questionnaire only.

Medical records of patients are reviewed to obtain information on pathological diagnosis and laboratory number, date of diagnosis, stage of disease, performance status, co-morbidities, and treatment plan. Medical records of partners may also be reviewed to obtain information on the incidence of smoking-related malignancies (i.e., cancer of the lung, larynx, esophagus, stomach, bladder, or head and neck).

Patients and their partners and first-degree relatives undergo blood sample collection for laboratory studies. Previously collected tumor samples are obtained from patients. Plasma DNA, lymphocyte DNA, and tumor DNA are analyzed by polymerase chain reaction (PCR) to identify loss of heterozygosity (LOH) between genomic (lymphocyte) DNA and the tumor and plasma DNA. Specific tumor-associated mutations are also analyzed by real-time PCR. Single nucleotide polymorphism studies, including common gene polymorphisms (metabolic genes, DNA repair genes, and tumor suppressor genes), in lung cancer families are also conducted.

A statistical model will be developed for future analysis and will include correlations in genetic alterations in DNA isolated from tumor and plasma, familial aggregation studies, and genetic analysis studies.

PROJECTED ACCRUAL: A total of 2,000 participants (500 patients and 1,500 partners and first-degree relatives [controls]) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient meeting the following criteria:

  * Pathologically confirmed lung cancer or planning to undergo lung cancer surgery pending pathological confirmation
  * Evidence of active disease (i.e., not in remission)
  * Meets 1 of the following criteria:

    * 60 years of age and under
    * Has a first-degree relative with lung cancer who is 60 years of age and under
    * Has two or more first- or second-degree relatives with lung cancer at any age
* Control meeting the following criteria:

  * Co-habiting partner of patient OR first-degree relative of patient or their partner
  * 18 years of age and over
* Resides within the North Trent Cancer Network region

PATIENT CHARACTERISTICS:

* Able and willing to complete study procedures

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Establishment of a resource bank of high quality genomic and plasma DNA and tumor and serum samples

SECONDARY OUTCOMES:
Analysis of single nucleotide polymorphisms for candidate lung cancer susceptibility genes in genomic DNA samples
Genetic changes of lung cancer in plasma DNA samples

CONTACTS AND LOCATIONS:
Overall Officials: Penella J. Woll, MD, PhD, Principal Investigator — Cancer Research Centre at Weston Park Hospital
Locations (1):
- Cancer Research Centre at Weston Park Hospital, Sheffield, England, United Kingdom